CLINICAL TRIAL: NCT05940675
Title: Generation Healthy Kids: A Cluster-randomized Trial of a Multi-component, Multi-setting Intervention to Promote Healthy Weight and Wellbeing in Danish School-aged Children
Brief Title: Generation Healthy Kids: A Cluster-randomized Trial of a Multi-component, Multi-setting Intervention
Acronym: GHK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: University of Southern Denmark (Other); Region Capital Denmark (Other); The Novo Nordisk Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: S-20220094
Record Dates: First submitted 2023-07-04; First posted 2023-07-11 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Childhood Obesity; Well-Being, Psychological; Physical Inactivity; Sleep; Screen Time; Diet Habit
Keywords: Obesity; Well-being; Physical activity; Sleep; Screen time; Community intervention; Socioeconomic Disparities in Health; Diet
MeSH Terms: conditions — Pediatric Obesity; Psychological Well-Being; Sedentary Behavior; Feeding Behavior; Obesity; Motor Activity | interventions — Food; Nutritional Status; Exercise; Sleep

STUDY DESIGN:
Intervention Model Description: 1:1
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Generation Healthy Kids intervention (Experimental): The intervention focuses on food and nutrition, physical activity, sleep and screen media habits, and engagement of the local stakeholders.
  Interventions: Behavioral: Food and Nutrition; Behavioral: Physical Activity (FitFirst); Behavioral: Sleep and screen media; Behavioral: Community capacity building
- Control (No Intervention): The schools will continue with their regular school schedules.

INTERVENTIONS:
Behavioral: Food and Nutrition — A key element is that children receive a free of charge healthy do-it-yourself school lunch 4 days per week. The meals adhere to the Nordic Nutrition Recommendations and the Danish Food-Based Dietary Guidelines with focus on fish, wholegrains, fruits and vegetables and drinking water as well as stimulation of children's food literacy. Other intervention components involve the after school clubs, local retail stores and the parents.
  Arms: Generation Healthy Kids intervention
Behavioral: Physical Activity (FitFirst) — To ensure that all children reach the recommended 3x30 minutes of vigorous activity per week, we will implement three weekly 40-minute sessions in the school curriculum. These sessions will be carried out throughout the study period and will encompass modified and varied sporting activities and games, which promote motivation, physical literacy, active involvement of all children, and high training intensity.
  Arms: Generation Healthy Kids intervention
Behavioral: Sleep and screen media — The aim of this component is to promote healthy sleep and screen media behaviours. Sleep and screen media recommendations will be presented for parents at three parent workshops and in electronic infographics. Teachers/pedagogues will facilitate small assignments on screen media and sleep practices with children during school time. Children will talk about and reflect upon screen media and sleep practices in their family, based on assignments and material from e.g., Medierådet (The Danish Media Council). The results of the children's assignments will be presented to their parents at later workshops. This is done to integrate the children's perspective in the parent workshops, especially in relation to screen media habits.
  Arms: Generation Healthy Kids intervention
Behavioral: Community capacity building — Community capacity building in selected local communities. To promote healthier eating, children and families need to be supported within their local community by food environments that make the healthy choice the easy choice and not a challenge in their everyday life. To promote physical activity, the children will be invited to participate in activities in the local sports clubs including camps in the holidays.
  Arms: Generation Healthy Kids intervention

SUMMARY:
The GHK intervention was developed according to the United Kingdom Medical Research Council's framework for developing and evaluating complex interventions. A pilot- and feasibility study was conducted during December 2022-April 2023, and the intervention was subsequently adapted and adjusted.

The GHK main trial is a two-school-year cluster-randomized school- and community trial designed to investigate the effect of the multi-setting, multi-component GHK intervention program on weight development, health and wellbeing in Danish children aged 6-11 years. The trial will include 24 schools in Denmark (12 intervention and 12 control).

The primary aim of the cluster-randomized trial is to investigate whether the GHK intervention program can promote healthy body composition as measured by fat mass (FM) in the intervention group compared with the control group. We hypothesize that the intervention will result in less FM gain in the intervention group compared with the control group over the two school-year study period.

DETAILED DESCRIPTION:
Generation Healthy Kids is a cluster-randomized school and community trial in which 24 schools will be randomly allocated to intervention or control. Schools are evenly distributed in two areas of Denmark: DK-EAST (Capital Region of Denmark and Region Zealand) and DK-WEST (Region of Southern Denmark). The overall study objective is to investigate if a 2-school-year multi-setting, multi-component intervention focusing on healthy diets, physical activity, sleep and screen media habits in the school and local community can promote healthy weight and body composition in children who are in 1st and 2nd grade at inclusion (i.e., age 6-9 years at inclusion). We will also investigate the intervention's effects on dietary intake and nutritional status; food literacy; family- and school meal culture, physical literacy, activity levels, and fitness; sleep and screen media habits; growth; cardio metabolic health; cognitive and motor functions; school performance; and mental health and well-being. Furthermore, we will evaluate the context, implementation and working mechanisms of the intervention.

In continuation of the above, we will investigate if the intervention can reduce social inequality in the outcomes, as well as explore potential effect modifiers such as sex, ethnicity, implementation levels, genetics, epigenetics etc. We will also explore associations between sociodemographic characteristics, health behaviors and outcomes cross-sectionally and longitudinally and use these data to validate and compare relevant measurement tools.

The innovative aspects of the Generation Healthy Kids study are the combination of an intervention targeting several important risk factors for excessive weight gain (dietary habits, physical activity, sleep, and screen time) with community capacity building and a systems approach. The unique combination is closely monitored for effect as well as process. The integrated intervention program will be distinctive in combining already tested effective intervention strategies with intervention components developed using co-creation and a systems mapping and working in varying settings of the child's life. Systems thinking will furthermore be used to ensure that a health equity lens is employed to understand the relationship between obesity and health inequalities locally. To reach children and families with low socio-economic status, focus will be on developing interventions that make healthy choices easy by creating healthy environments around the children, both at school and during leisure time.

ELIGIBILITY:
Inclusion Criteria:

* All children attending 1st or 2nd grade in the recruited schools

Exclusion Criteria:

- No exclusion criteria will be applied. If parents, teachers or research staff judge that a child cannot participate in certain parts of the intervention or measurement schedule, e.g. due to severe allergies, chronic diseases or mental/physical disabilities, the child will be eligible to participate in the remaining parts of the study.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1372 (Actual)
Dates: Start 2023-08-14 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Fat mass in kg | Baseline and 18-20 months
  Between group difference in change in fat mass measured by bioimpedance analysis (InBody 270).

SECONDARY OUTCOMES:
Fat mass in kg (2) | Baseline , 6-8 months, 18-20 months
  Between group difference in change in fat mass measured by a bioimpedance analysis (InBody 270).
Fat free mass in kg | Baseline , 6-8 months, 18-20 months
  Between group difference in change in fat free mass measured by a bioimpedance analysis (InBody 270).
Fat mass index in kg/m2 | Baseline , 6-8 months, 18-20 months
  Between group difference in change in fat mass index measured by a bioimpedance analysis (InBody 270).
Fat free mass index in kg/m2 | Baseline , 6-8 months, 18-20 months
  Between group difference in change in fat free mass index measured by a bioimpedance analysis (InBody 270).
Fat-Free-Mass-to-Fat-Mass ratio | Baseline , 6-8 months, 18-20 months
  Between group difference in change in FFM-to-FM ratio measured by a bioimpedance analysis (InBody 270).
% Fat Mass | Baseline , 6-8 months, 18-20 months
  Between group difference in change in % FM in kg measured by a bioimpedance analysis (InBody 270).
Height in cm | Baseline , 6-8 months, 18-20 months
  Between group difference in change in standing height measured using a portable stadiometer.
Weight status in % | Baseline , 6-8 months, 18-20 months
  Between group difference in change in prevalence of children with underweight, normalweight, overweight and obesity, based on the cutoffs defined by Cole et al. and the International Task Force of Obesity. Body weight is measured by a bioimpedance analysis (InBody 270) and height by using a portable stadiometer.
BMI z-score | Baseline , 6-8 months, 18-20 months
  Between group difference in change in BMI z-score based on WHO references. Weight and height is measured using weight from the bioimpedance analysis (InBody 270) and a portable stadiometer, respectively.
Waist circumference in mm | Baseline , 6-8 months, 18-20 months
  Between group difference in change in waist circumference to the nearest mm by a non-elastic measuring tape at the level of the umbilicus.

OTHER OUTCOMES:
Health related quality of life | Baseline , 6-8 months, 18-20 months
  Between group difference in change in the total summary score of health-related quality of life measured with the KIDSCREEN 27 child self-report questionnaire. Data is collected using an adapted video and speech assisted electronic version with a smiley scale for each answer. The questionnaire assesses the child's physical well-being (5 items), psychological well-being (7 items), autonomy and parent relation (7 items), peers and social support (4 items), and school environment (4 items).
Mental health | Baseline , 6-8 months, 18-20 months
  Between group difference in change in the total difficulties score of the Strengths and difficulties questionnaire. Assessed using the parent-reported version of the Strengths and Difficulties Questionnaire. An overall total difficulties score is calculated, along with five subscale scores: emotional symptoms, conduct problems, hyperactivity/Inattention, relationship problems, and prosocial behavior.
Resting blood pressure in mmHg | Baseline , 6-8 months, 18-20 months
  Between group difference in change in systolic and diastolic blood pressure.
Resting heart rate beats/min | Baseline , 6-8 months, 18-20 months
  Between group difference in change in heart rate.
Plasma lipid profile in mmol/L | Baseline and 6-8 months, (18-20 months if funding is available)
  Between group difference in change in plasma total, LDL and HDL cholesterol and triacylglycerol. Only among children in DK-EAST.
Plasma insulin in pmol/L. | Baseline and 6-8 months, (18-20 months if funding is available)
  Between group difference in change in plasma insulin. Only among children in DK-EAST.
Plasma glucose in mmol/L. | Baseline and 6-8 months, (18-20 months if funding is available)
  Between group difference in change in plasma glucose. Only among children in DK-EAST.
Aerobic fitness and intermittent exercise performance | Baseline, 6-8 months, 18-20 months
  Between group difference in change in aerobic fitness and intermittent exercise performance.
Sprint performance | Baseline, 6-8 months, 18-20 months
  Between group difference in change in sprint performance as measured by 20 m sprint test.
Muscular fitness and strength | Baseline, 6-8 months, 18-20 months
  Between group difference in change in muscular fitness and strength.
Balance ability | Baseline and 18-20 months
  Between group difference in change in balance ability.
Jump height | Baseline and 18-20 months
  Between group difference in change in jump height (countermovement jump).
Upper and lower extremity gross motor function | Baseline and 18-20 months
  Between group difference in change in Upper and lower extremity gross motor function.
Agility | Baseline and 18-20 months
  Between group difference in change in agility will be assessed using the Canadian Exercise and Movement Skills Assessment (CAMSA)
Physically active behavior | Baseline, 18-20 months
  Between group change in total time spent being physical active. Non-sedentary time is defined as any waking activity characterized as not being in a sitting, reclining or lying posture with minimal stationary movement. Activity is measured for 7 consecutive days using a thigh worn accelerometer (Axivity AX3).
Moderate to vigorous physical activity | Baseline, 18-20 months
  Between group change in time spent in moderate to vigorous physical activity. Moderate to vigorous physical activity is measured for 7 consecutive days using a thigh worn accelerometer (Axivity AX3).
Total sleep time | Baseline, 18-20 months
  Between group change in total sleep time. Sleep is measured for 7 consecutive days using a thigh worn accelerometer (Axivity AX3).
Sleep quality | Baseline , 6-8 months, 18-20 months
  Between group difference in change in sleep quality, as measured by Child Sleep Habits Questionnaire (parent-reported).
Total screen time | Baseline , 6-8 months, 18-20 months
  Between group difference in change in total screen time (hours), as measured by modified SCREENS questionnaire (parent-reported).
Smartphone and tablet usage | Baseline , 6-8 months, 18-20 months
  Between group difference in change in smartphone/tablet usage, objectively assessed over 14 days using Ethica application.
Food literacy | Baseline, 6-8 months, 18-20 months
  Between group difference in change in child-reported using a GHK food literacy and meal culture questionnaire currently under development
School meal culture | Baseline, 6-8 months, 18-20 months
  Between group difference in change in child-reported using a GHK food literacy and meal culture questionnaire currently under development
Family meal culture | Baseline, 6-8 months, 18-20 months
  Between group difference in change in child-reported using a GHK food literacy and meal culture questionnaire currently under development
Dietary intake in g/day | Baseline, 6-8 months, 18-20 months
  Between group difference in change in dietary intake by 3-day electronic dietary record and FFQ.
n-3 long-chain polyunsaturated fatty acid (LCPUFA) status in weight% | Baseline and 6-8 months, (18-20 months if funding is available)
  Between group difference change in wholeblood n-3 LCPUFA status (eicosapentaenoic acid and docosahexaenoic acid). Only among children in DK-EAST.
Blood hemoglobin in mmol/L. | Baseline and 6-8 months, (18-20 months if funding is available)
  Between group difference in change in wholeblood hemoglobin (iron status). Only among children in DK-EAST.
Serum ferritin in ug/L. | Baseline and 6-8 months, (18-20 months if funding is available)
  Between group difference in change in serum ferritin (iron status). Only among children in DK-EAST.
Serum 25-hydroxyvitamin D in nmol/L. | Baseline and 6-8 months, (18-20 months if funding is available)
  Between group difference in change in serum 25-hydroxyvitamin D (vitamin D status). Only among children in DK-EAST.
Insulin-like growth factor-1 in ug/L. | Baseline and 6-8 months, (18-20 months if funding is available)
  Between group difference in change in serum insulin-like growth factor-1 (growth factor). Only among children in DK-EAST.
Processing speed | Baseline and 18-20 months
  Performance in neuropsychological assessment of processing speed as choice reaction time (Cambridge Neuropsychological Test Automated Battery, Cambridge cognition, UK).
Sustained attention | Baseline and 18-20 months
  Performance in neuropsychological assessment of sustained attention ability assessed as errors during a sustained test procedure (Cambridge Neuropsychological Test Automated Battery, Cambridge cognition, UK).
Spatial working memory | Baseline and 18-20 months
  Performance in neuropsychological assessment of spatial working memory assessed as errors and strategy during the test procedure (Cambridge Neuropsychological Test Automated Battery, Cambridge cognition, UK).
Inhibitory control | Baseline and 18-20 months
  Performance in neuropsychological assessment of inhibitory control assessed as errors during the test procedure (Cambridge Neuropsychological Test Automated Battery, Cambridge cognition, UK).
Cognitive flexibility | Baseline and 18-20 months
  Performance in neuropsychological assessment of cognitive flexibility assessed as errors during the test procedure (Cambridge Neuropsychological Test Automated Battery, Cambridge cognition, UK).
Fine motor control | Baseline and 18-20 months
  Performance in neuropsychological assessment of fine motor control assessed as endpoint accuracy during the test procedure (Cambridge Neuropsychological Test Automated Battery, Cambridge cognition, UK).
School performance - Danish reading comprehension | Baseline and 18-20 months
  Between group difference in change in Danish reading skills (Hogrefe, Denmark).
School performance - mathematics proficiency | Baseline and 18-20 months
  Between group difference in change in mathematics proficiency (Hogrefe, Denmark).
School absence due to sickness and other causes | Baseline, 6-8 months, 18-20 months
  Between group difference in change in number of days abscent from school due to sickness recorded in school registration data
Physical literacy | Baseline, 18-20 months
  Between group difference in change in total score of physical literacy as well as for the emotional, cognitive and physical subdomain

CONTACTS AND LOCATIONS:
Overall Officials: Nikolai B Nordsborg, PhD, Study Director — University of Copenhagen; Jens Troelsen, PhD, Principal Investigator — University of Southern Denmark; Ulla Toft, PhD, Study Chair — Capitol Region of Southern Denmark
Locations (2):
- Denmark (2):
  - 11 schools in the Capital Region of Denmark and Region Zealand, Copenhagen, Capital Region and Region Zealand
  - 12 Schools in Region of Southern Denmark, Odense, Region Syddanmark

IPD SHARING:
Plan to Share IPD: Yes
Only de-indentified data will be shared.
Supporting Information: Study Protocol, SAP
Access Criteria: A formal application must be approved by the study's steering committee.

REFERENCES:
- [Derived] Thomsen LT, Schmidt-Persson J, Damsgaard CT, Krustrup P, Grontved A, Krolner RF, Nielsen G, Lundbye-Jensen J, Skovgaard T, Molgaard C, Hansen ABG, Hoeeg D, Larsen MN, Lund L, Melby PS, Pedersen NH, Troelsen J, Nordsborg NB, Toft U. Generation Healthy Kids: Protocol for a cluster-randomized controlled trial of a multi-component and multi-setting intervention to promote healthy weight and wellbeing in 6-11-year-old children in Denmark. PLoS One. 2024 Dec 5;19(12):e0308142. doi: 10.1371/journal.pone.0308142. eCollection 2024. PMID 39636875

DOCUMENTS (8):
  • Study Protocol: Version 1.1, 6 March 2023 (2023-03-06): https://cdn.clinicaltrials.gov/large-docs/75/NCT05940675/Prot_000.pdf
  • Study Protocol: Version 3.0, 25 July 2023 (2023-07-25): https://cdn.clinicaltrials.gov/large-docs/75/NCT05940675/Prot_002.pdf
  • Study Protocol: Version 4.0, 26 February 2024 (2024-02-26): https://cdn.clinicaltrials.gov/large-docs/75/NCT05940675/Prot_003.pdf
  • Study Protocol: Version 5.0, 7 November 2024 (2024-11-07): https://cdn.clinicaltrials.gov/large-docs/75/NCT05940675/Prot_004.pdf
  • Study Protocol: Version 6.0, 17 January 2025 (2025-01-17): https://cdn.clinicaltrials.gov/large-docs/75/NCT05940675/Prot_005.pdf
  • Study Protocol: Version 2.2, 10 July 2023 (2023-07-10): https://cdn.clinicaltrials.gov/large-docs/75/NCT05940675/Prot_007.pdf
  • Statistical Analysis Plan: Version 1.0, dated 11 June 2025 (2025-06-11): https://cdn.clinicaltrials.gov/large-docs/75/NCT05940675/SAP_008.pdf
  • Statistical Analysis Plan: Version 2.0, dated 18 November 2025 (2025-11-18): https://cdn.clinicaltrials.gov/large-docs/75/NCT05940675/SAP_009.pdf